CLINICAL TRIAL: NCT05685628
Title: Evaluation of the Quality of Life Induced by the Cinnamon Anti-odor Dressing in Patients With Malodorous Wounds: a Multicenter Randomized Controlled Trial
Brief Title: Evaluation of the Quality of Life Induced by the Cinnamon Anti-odor Dressing in Patients With Malodorous Wounds
Acronym: CINNAMON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP220093
Record Dates: First submitted 2022-12-07; First posted 2023-01-17 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Malodorous Wounds (Chronic, Malignant or Infected Wounds)
Keywords: Malodorous wounds; Malignant wound; Symptom management
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cinnamon dressing group (Experimental): Use of the cinnamon dressing for 14 days
  Interventions: Other: Cinnamon dressing
- Charcoal dressing Group (Active Comparator): Use of the charcoal dressing for 14 days
  Interventions: Other: Charcoal dressing

INTERVENTIONS:
Other: Cinnamon dressing — Use of CINESTEAM® as a non-occlusive secondary dressing
  CE marked medical device class I, secondary, absorbent, non-adhesive and composed of:
  * Anti-odor upper part, adsorbent containing cinnamon powder.
  * Weakly absorbent lower part intended to absorb excess exudates.
  Arms: Cinnamon dressing group
Other: Charcoal dressing — Use of a secondary non-occlusive activated charcoal dressing (brand of your choice)
  Arms: Charcoal dressing Group

SUMMARY:
Refer to "Detailed description".

DETAILED DESCRIPTION:
Wounds can smell bad when they are necrotic, infected, malignant or complicated by fistulas or abscesses. The discomfort and evocations (perception) associated with these smells can be different from person to person. Foul odors are often associated with a repulsive effect. Malodorous wounds can have negative social and psychological repercussions (shame, depreciation, isolation).

Malodor is due to the presence of bacteria, whether the wound is colonized or infected. Bacteria release Volatile Organic Compounds (VOCs) that emit these odors. There are a multitude of anti-odor treatments (conventional or not) that highlight the difficulty of effectively treating this symptom.

Charcoal dressings are recommended. Charcoal does not treat the etiology, it is not odorous, but it has the ability to adsorb VOCs.

To treat odor, the most prescribed antibiotic is Metronidazole, because its action targets anaerobic bacteria whose presence increases odor. But repeated prescriptions of antibiotics increase the risk of selection pressure, in addition to possible side effects. It's not efficient in all the situations

Another strategy is the application of local antimicrobials. But it is effective only if the bacteria responsible for the odors are on the surface of the wound, which is not the case if it is a tumor mass, thick necrosis or abscesses.

These local or general treatments do not completely control bad odors in all situations. A new dressing combining adsorption capabilities (reduction of bad odors) with odor release (modification of the perception of residual odors) with cinnamon (CINESTEAM®) is now available.

This work aims to evaluate this new medical device compared to the reference dressing (charcoal) on quality of life, as well as criteria still poorly documented such as discomfort and appetite.

The primary endpoint is the percentage of patients with a reduction of at least 0.4 points in the overall score on the Wound-Qol questionnaire (Quality of life). It is estimated that a 0.4 point reduction in the overall score is a clinically relevant reduction for patients and reflects an improvement in their quality of life. An improvement of 0.4 points is expected in 25% of patients in the control arm (charcoal dressing) and in 55% of patients in the experimental arm (cinnamon dressing).

The study provides for the inclusion of 98 people with malodorous wounds in several hospital located on Ile de France.

Day 0: General data on the wound and current treatments will collected, Wound-Qol scale, lifestyle, discomfort related to smell, evaluation of appetite. The evaluated dressings will positioned on the top of primary dressing. They will fix by a non-occlusive or semi-occlusive fixation. The entire dressing will changed 1 time a day for 14 days.

Day 1: The patient will assess the discomfort related to the smell before changing the dressing.

Day 3: Assessment of the employability of the dressing by the caregiver.

Day 7 and 14: Assessment of the discomfort related to the smell by the patient, the caregiver and the entourage. Appetite will assessed with the Simple Evaluation of Food Intake scale (SEFI). Day 14 only: Wound-Qol scale and self-questionnaire on the appearance of any discomfort(s)/reaction(s) due to the dressing.

ELIGIBILITY:
Inclusion Criteria:

* Patient >18 years of age with a smelly wound (discomfort > 4/10 expressed by the patient);
* Predictive wound healing >14 days (clinical judgement);
* Patient benefiting from a social security scheme (AME excluded)
* Patient, and curator if applicable, informed and having signed the consent form for participation in the study

Exclusion Criteria:

* Patient already receiving a secondary charcoal or cinnamon dressing
* Patient with pressure ulcer stage 1 or 2
* Patient treated by metronidazole or antimicrobial for < 3 days;
* Patient who cannot communicate his feelings;
* Anosmic patient;
* Patient with cinnamon allergy;
* Persons deprived of their liberty or under guardianship;
* Inability to submit to the medical follow-up of the trial for geographical, social, psychological or cognitive reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2027-04-19 (Estimated); Study Completion 2027-04-19 (Estimated)

PRIMARY OUTCOMES:
Wound-Qol | Day 0 and 14
  Wound-QoL (Questionnaire on quality of life with chronic wounds) measures the disease-specific, health-related quality of life of patients with chronic wounds. It can be used in clinical and observational studies as well as in daily practice. Two versions are available and we decided to use the original version (Wound-QoL-17) with 17 items. The primary endpoint is the reduction of more than 0.4 points in the overall score of the Wound-Qol quality of life questionnaire between D0 and D14.

SECONDARY OUTCOMES:
Odor discomfort / patient | Day 0, 7 and 14.
  Discomfort related to the smell felt in the last 24 hours (from 0 to 10) assessed by the patient.
Odor discomfort / nurse | Day 0, 7 and 14.
  Discomfort related to the smell felt (from 0 to 10) assessed by the nurse performing the treatment
Odor discomfort / family | Day 0, 7 and 14.
  Discomfort related to the smell felt (from 0 to 10) assessed by the family present (if it's practical)
SEFI® Scale to assess appetite | Day 0, 7 and 14.
  SEFI® is a quick and simple tool of assessment of food intake and consists in a visual analogue scale (0 to 10), or evaluation of consumed portions
Odor discomfort / patient | Day 1
  Discomfort related to the smell felt (from 0 to 10) assessed by the patient just before the first dressing change
Cutaneous reaction or dressing discomfort | Day 14
  Patient's questionnaire
Dressing qualities | Day 3
  Nurse's questionnaire: dressing flexibility, application, opening

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle FROMANTIN, IDE, Study Director — Institut Curie
Locations (6):
- France (6):
  - Hôpital Henri Mondor, Créteil
  - Hospitalisation à domicile Fondation Santé Service, Levallois-Perret
  - Hospitalisation à Domicile AP-HP, Paris
  - Institut Curie, Paris
  - Hôpital Saint Louis, Paris
  - Hôpital Sainte Périne, Paris

IPD SHARING:
Plan to Share IPD: No
Data are own by Assistance Publique - Hôpitaux de Paris, please contact sponsor for further information.